CLINICAL TRIAL: NCT05413993
Title: Immediate Effect Of Photobiomodulation On Ph And Salivary Flow: Quasi-Experimental Clinical Trial
Brief Title: Effect of Photobiomodulation on ph and Salivary Flow
Acronym: PBMSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD, University of Nove de Julho
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBMSF
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Xerostomia
Keywords: saliva flow; photobiomodulation
MeSH Terms: conditions — Xerostomia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: QUASI-EXPERIMENTAL CLINICAL TRIAL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra and extraoral application (Active Comparator): The laser was applied for 60 seconds, in 2 intraoral points and 2 extraoral points.
  Interventions: Radiation: photobiomodulation
- extraoral application (Experimental): The laser was applied only extraoral points
  Interventions: Radiation: photobiomodulation

INTERVENTIONS:
Radiation: photobiomodulation — Laser application intraorals and extraoral points in the region of the salivary glands bilaterally

SUMMARY:
Changes in salivary parameters, such as decreased flow, changes in pH and composition, can lead to changes in oral health. Saliva is responsible for the homeostasis of the oral cavity and is therefore directly related to the occurrence of caries, periodontitis, fungal and bacterial infections. These situations compromise the quality of life of the population and for this reason prevention and treatment strategies need to be studied and developed. Photobiomodulation is an alternative that has been increasingly practiced by health professionals. It consists of the application of light to a biological system that is capable of inducing a photochemical process, mainly in the mitochondria, thus stimulating the production of energy in the form of adenosine triphosphate (ATP), which can increase cellular metabolism and produce effects. as analgesia and tissue regeneration. In dentistry, studies using photobiomodulation have shown promise in improving some salivary parameters. This study aimed to compare the action of infrared light on salivary flow and pH, using two application techniques: extraoral (G1) and intra and extraoral (G2), with the application interval between the two techniques being 7 days

DETAILED DESCRIPTION:
This is a quasi-experimental clinical study evaluating the flow and salivary pH of healthy adults. The study was carried out with 20 adult patients at the Nove de Julho University. This study aimed to compare the action of infrared light on salivary flow and pH, using two application techniques: extraoral (G1) and intra and extraoral (G2), with the application interval between the two techniques being 7 days. The sample consisted of 20 healthy adults, who participated in both groups, thus being the actual control in the evaluations. Stimulated saliva was collected in both groups before and immediately after light application. In G1, a cluster with 3 spots was used, at a wavelength of 808 nanometers, power of 120 mW, with 24J of energy on the extraoral surface, for 67 seconds, in the region of the parotid gland, region of the submandibular and sublingual glands bilaterally, totaling 4 application regions, with total deposited energy of 96 joules. In G2, the laser was applied for 60 seconds, in 2 intraoral and 2 extraoral points in the region of the parotid glands bilaterally, as well as 1 intraoral and 1 extraoral point in the regions of the submandibular and sublingual glands (totaling 16 points), with a central wavelength of 808 nm; continuous operating mode; power of 100mW; with an aperture diameter of 0.354 cm (with spacer); radiant energy of 6J per point, totaling 96 joules of energy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over 18 years of age
* healthy dentition.

Exclusion Criteria:

* dental caries
* gingivitis or other alterations in the oral cavity
* who use medication that has the side effect of decreasing the salivary flow,
* who have used an antibiotic or anti-inflammatory within the last 30 days,
* diabetes.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change in salivary flow | 30 minutes
  The saliva was collected at the Dental Clinic of the Universidade Nove de Julho, with the adult seated at the dental team. To obtain the stimulated saliva, we used sialogogue chewing for 5 minutes, and the saliva collection was performed, by expectoration of all the saliva accumulated in the mouth every 1 minute of chewing, inside graduated glass tubes. Stimulated saliva was collected before and immediately after laser application. This procedure is performed both in the extraoral application only, and in the intra and extraoral application. After collection, 3 drops of simethicone were used to eliminate gases and foam, and only after this procedure the volume of saliva collected was measured.

SECONDARY OUTCOMES:
Change in pH salivary | 30 minutes
  The saliva tube was properly placed on a bench for immediate pH measurement with a colorimetric tape (MERCK Ⓡ Quimical, São Paulo, Brazil) inside the collecting device. The tape features a pH scale from 0 to 14.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho Univ, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No